CLINICAL TRIAL: NCT06232681
Title: The Effect of Progressive Relaxation Exercises Applied to Family Members Caregiving for Hemiplegic Patients on Caregiving Burden and Meaning of Life
Brief Title: The Effect of Progressive Relaxation Exercises Applied to Caregivers on Caregiving Burden and Meaning of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: kıvan çevik kaya (Other)
Responsible Party: Sponsor-Investigator, kıvan çevik kaya, Celal Bayar University, Celal Bayar University
Organization: Celal Bayar University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MCBU-K-CEVIK-003
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Hemiplegia
Keywords: progressive relaxation exercise; burden; caregiver; the meaning of life
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive relaxation exercise application (Experimental): Progressive relaxation exercise practice Those who agree to participate in the study will be asked to fill in the Patient and Patient Relative Form, Cheltanhams Patient Classification Scale, Caregiving Burden Scale and Meaning and Purpose of Life Scale, which include personal information and information about the patient. Relaxation exercises will be explained and demonstrated by the researcher (Funda AKTÜRK) once a day for 1 month starting from the hospitalisation to the clinic and will be played on the computer. You will be asked to perform these exercises after listening to the video (CD). Relaxation exercises are exercises based on stretching and relaxing your muscles. Before the application, in the middle of the application (15th day) and at the end of the application, all forms except the introduction form will be filled in again.
  Interventions: Behavioral: Progressive relaxation exercise
- Control group (No Intervention): The participants in the control group also filled in the data collection tools without undergoing any intervention.

INTERVENTIONS:
Behavioral: Progressive relaxation exercise — The intervention group will take one month progressive relaxation exercise starting from the hospitalisation to the clinic
  Arms: Progressive relaxation exercise application

SUMMARY:
This randomised controlled experimental type study will be conducted with family members who care for the relatives of hemiplegic patients who are hospitalised in Manisa Merkezefendi and Turgutlu State Hospital Physical Therapy Services.

DETAILED DESCRIPTION:
The population of the study will consist of the caregivers of hemiplegic patients receiving treatment in the clinic on the specified dates in Turgutlu State Hospital and Manisa Merkezefendi State Hospital Physical Therapy Service. The sample will consist of individuals who meet the inclusion criteria. Individuals in Turgutlu State Hospital will constitute the intervention group of the study and individuals in Manisa Merkezefendi State Hospital will constitute the control group of the study. The aim of this study was to determine the effect of progressive relaxation exercises applied to family members caring for hemiplegic patients on caregiving burden and meaning of life. In the intervention group, those who agree to participate in the study will be asked to fill in the Patient and Patient Relative Form, Cheltanhams Patient Classification Scale, Caregiving Burden Scale and Meaning and Purpose of Life Scale, which include personal information and information about the patient. Relaxation exercises will be explained and demonstrated by the researcher (Funda AKTÜRK) once a day for 1 month starting from the hospitalisation to the clinic and will be played on the computer. You will be asked to perform these exercises after listening to the video (CD). Relaxation exercises are exercises based on stretching and relaxing your muscles. Before the application, in the middle of the application (15th day) and at the end of the application, all forms except the introduction form will be filled in again. In the Control Group, those who agree to participate in the study will be asked to fill in the;Patient and Patient Relative Form, Cheltanhams Patient Classification Scale, Caregiving Burden Scale and Meaning and Purpose of Life Scale, which include personal information and information about the patient. The control group will be asked to fill in the forms at the same time as the intervention group without any intervention. If requested, progressive relaxation exercises will be applied to the control group after the end of the study

ELIGIBILITY:
Inclusion Criteria:

* Family members who have no communication problems,
* Who are 18 years of age or older,
* Whose patient will be hospitalised in the clinic for at least one month,
* Who agree to participate in the study will be recruited.

Exclusion Criteria:

* Individuals who have communication problems,
* The caregiver is not a family member,
* are 18 years of age or younger,
* The patient stays in the clinic for less than one month,
* Has previously received progressive relaxation training, and who do not agree to participate in the study will be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2024-04-19 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Care burden | 30 day
  Caregiving Burden Scale was used. The scale has a Likert-type evaluation ranging from 0 to 4 in the form of never, rarely, sometimes, frequently, often, or almost always. A minimum score of 0 and a maximum score of 88 can be obtained from the scale. The items in the scale are generally related to the social and emotional domain, and a high scale score indicates that the distress experienced is high.
The meaning and purpose of life | 30 day
  Meaning and Purpose of Life Scale was used. The Life's Meaning and Purpose Scale, which is prepared in Likert style and answered by marking one of the options of strongly agree, agree, undecided, disagree and strongly disagree according to frequency, consists of a total of (17) items including (11) positive and (6) negative statements. The options ticked for positive statements are evaluated by scoring as strongly agree (5), agree (4), undecided (3), disagree (2) and strongly disagree (1) respectively, while the options ticked for negative statements are evaluated by scoring in reverse order as strongly agree (1), agree (2), undecided (3), disagree (4) and strongly disagree (5). The lowest score that can be obtained from the scale is (17x1=17) and the highest score is (17x5=85). A high score indicates a high level of meaning in individuals' lives, while a low score indicates a low level of meaning.

CONTACTS AND LOCATIONS:
Overall Officials: Funda AKTÜRK, Principal Investigator — Celal Bayar University
Locations (1):
- Manisa Celal Bayar University, Manisa, Yunusemre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data will be given if it's necessary and if it is not problem for ethical office.